CLINICAL TRIAL: NCT06376110
Title: A Split-Face, Single-Blind, Study Assessing the Use of a Topical Antioxidant Containing Silymarin With A Series of 1726nm Laser Procedures to Reduce Sebum Production
Brief Title: Single-Blind Study Assessing the Use of a Topical Antioxidant With A Series of Laser Procedures to Reduce Sebum Production
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Austin Institute for Clinical Research (Network)
Collaborators: SkinCeuticals (Unknown)
Responsible Party: Principal Investigator, Edward Lain, MD, Principal Investigator, Austin Institute for Clinical Research
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: AviClear-001
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Topical Antioxidant Serum containing Silymarin CF (Left Face) (Active Comparator): 14 day application of topical antioxidant serum containing Silymarin CF
  Subjects will be given study drug and instructed to topically apply to the treatment area, the respectively randomized half of the face, once daily for 14 consecutive days.
  Interventions: Drug: Topical Antioxidant Serum; Device: AviClear Laser
- Topical Antioxidant Serum containing Silymarin CF (Right Face) (Active Comparator): 14 day application of topical antioxidant serum containing Silymarin CF
  Subjects will be given study drug and instructed to topically apply to the treatment area, the respectively randomized half of the face, once daily for 14 consecutive days.
  Interventions: Drug: Topical Antioxidant Serum; Device: AviClear Laser

INTERVENTIONS:
Drug: Topical Antioxidant Serum — An oil-free vitamin C serum for oily skin and blemish-prone skin that delivers advanced environmental protection, reduces oiliness, refines skin texture, and visibly improves skin clarity and fine lines.
  Other Names: SkinCeuticals Silymarin CF
Device: AviClear Laser — The AviClear (1726nm) laser is FDA-cleared for use on mild to severe inflammatory acne, with a recommended treatment course comprised of 3 laser procedures each one month apart.

SUMMARY:
This is a split-face, single-blind study assessing the use of an antioxidant serum with a series of acne laser treatments to reduce sebum production in healthy male and female subjects between the ages of 18 and 65 years, inclusive, with Fitzpatrick skin types I-VI.

DETAILED DESCRIPTION:
A single-center study. Clinical efficacy will be assessed using Investigator Global Assessment (IGA). Instrumentation will be assessed using VISIA imaging procedures, and sebumeter (sebum production). Tolerability will be assessed in subjects through objective tolerance grading and subjective tolerance assessment. In addition, subject perception of product will be evaluated by questionnaires. Live investigator clinical efficacy grading, tolerance evaluations, and subject self-assessments; will be performed at baseline (Day 0), Day 14, Day 42, and Day 70. Additionally instrumentation measurements of erythema and hyperpigmentation will be calculated by digital assessments of facial photographs.

All data will be collected by the clinical site and delivered to SGS in Excel files, including demographic information, clinical grading of efficacy and tolerability evaluations, sebumeter, and self-assessment questionnaire data. Data review and analyses will be performed by an independent data committee. Interim topline data will be sent to the Sponsor after Day 14, 42, and 70. End-of-study topline data will be sent at 10 business days after study completion. A clinical study report will be drafted using an SGS report template and incorporating any documented Sponsor preferences on file with SGS. The draft report will be submitted to the Sponsor for approval prior to finalization, and revisions may be made at the Sponsor's request. SGS will submit the draft report to the Sponsor 20-30 business days after approval of al statistical analysis and receipt of study documents from the study site. Any additions and changes to the statistical analysis after study completion may delay issuance of the draft report. After receiving the draft report, the Sponsor will have 6 months to make revisions. If SGS has received no revisions or comments within 6 months, the report will be approved for finalization. Every effort will be made to send the final report to the Sponsor within 10 business days after Sponsor approval or after the 6-month period has passed.

A total of 10 subjects are planned to be enrolled. Subjects who met the specified inclusion/exclusion criteria will be randomized to receive the topical antioxidant on one side and placebo on the other side on Day 0 of the study. On Day 14 of the study, each subject will receive the first acne laser treatment to the entire face. Additional laser treatments, and subject visits, occur on Days 42 and 70, with the final follow-up visit on Day 98. All evaluations will be done in a single-blind fashion. Clinical efficacy endpoints will be evaluated on Days 14, 42, 70, and 98. Tolerance endpoints will be evaluated on Days 0, 14, 42, and 70. Physician assessments, sebumeter readings, patient-reported outcomes, and photographs will be captured during this study.

A subject may be discontinued from study treatment at any time if the subject, the Investigator, or the Sponsor feels that it is not in the subject's best interest to continue. If a subject is withdrawn from treatment due to an AE, the subject will be followed and treated by the Investigator until the abnormal parameter or symptom has resolved or stabilized.

All subjects who discontinue study treatment should come in for an early discontinuation visit as soon as possible and then should be encouraged to complete all remaining scheduled visits and procedures. All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice. If a subject withdraws prior to or during the procedure, an additional subject may be enrolled to replace the withdrawn subject. The Sponsor may elect to close the trial at any time during the course of the study. Any data collected prior to termination may be analyzed as specified in the protocol.

The Investigator will probe, via discussion with the subject, for the occurrence of AEs (adverse events) during each subject visit and record the information in the site's source documents. Adverse events will be recorded in the subject CRF (case report form). Adverse events will be described by duration (start and stop dates and times), severity, outcome, treatment and relation to study drug, or if unrelated, the cause. The study site will document all SAEs (serious adverse events) that occur (whether or not related to study treatment). The collection period for all SAEs will begin after informed consent is obtained and end after procedures for the final study visit have been completed.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the inclusion criteria in order to be eligible for this study:

1. Healthy male and female subjects aged between 18 and 65 years, inclusive of all Fitzpatrick Skin Types (I-VI)
2. Self-perceived "oily skin". Subject must answer "Yes" to the question "Do you have an oily complexion?"
3. Mild to moderate acne (2-3) based on IGA
4. No known medical conditions that, in the Investigator's opinion may interfere with study participation
5. Female subjects of childbearing potential must be on and remain on a study-specified stable form of birth control throughout participation in study (See Section 6.1.1)
6. Willingness to cooperate and participate by following study requirements
7. Individuals must sign an informed consent and a photography consent

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Subjects that are being treated for cancer or have a history of facial skin cancer on the test areas
2. Subjects with sunburn, moderate to pronounced suntan, pronounced asymmetric skin aging, tattoos, scars or other disfiguration, dilated vessels or other conditions on the test area that might influence the test results
3. Subjects currently taking certain medications which in the opinion of the Investigators may interfere with the study. This includes but not limited to routine high dosage use of anti-inflammatory drugs (aspirin, ibuprofen, corticosteroids [steroid nose drops, inhalers and/or eye drops are permitted]), and immunosuppressive drugs
4. Subjects with self-reported, uncontrolled systemic disease which, in the opinion of the Investigator, may hinder either the subject 's ability to perform all responsibilities of the trial or the Investigator's ability to perform assessments
5. Females known to be pregnant, nursing or planning to become pregnant
6. Subjects participating in other facial clinical studies
7. Subjects who have routinely used an alpha-hydroxy-acid (AHA) or a beta-hydroxy-acid (BHA) containing product within two weeks or Retin-A, Retin-A Micro, Renova ,Differin , Avita, Tazorac, or Soriatane within 8 weeks of the study start or have taken Accutane within one year of the study start. Subjects who have used Retinol in the last 8 weeks
8. Subjects with history of severe acne flares
9. Subjects who have had ablative laser treatments, microneedling, and/or chemical peels or dermabrasion within the last six months
10. Subjects who have had non-ablative laser treatments or IPL within the last 3 months
11. Subjects with known allergies to skin treatment products or cosmetics, toiletries, and/or topical drugs
12. Subjects currently using topically applied prescription medications on the face

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Change in Facial Acne Severity | Change from Baseline at Day 98
  Measured by Live Clinical Investigator grading of overall severity of facial acne using the Investigator Global Assessment (IGA). The parameters of the scale are as follows, 0 = clear (best possible outcome), 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe (worst possible outcome). A decrease in scores indicates an improvement in study treatment efficacy. The null hypothesis is that the mean change from baseline is zero.
Change in Subject Tolerability | Change from Baseline at Day 98
  Measured by Live Clinical Investigator grading by subject reporting of burning, stinging, and itching. Each will be measured with the following parameters, 0 = none (best possible outcome), 1 = mild, 2 = moderate, and 3 = severe (worst possible outcome). A decrease in scores or lack of significant increases indicate tolerability of the study treatment. The null hypothesis is that the mean change from baseline is zero.

SECONDARY OUTCOMES:
Change in Skin Quality | Change from Baseline at Day 98
  Measured by Live Clinical Investigator Assessment of Redness, Skin Clarity, Appearance of Pores, Skin Texture/Smoothness (Visual), Skin Texture/Smoothness (Tactile), Hyperpigmentation, Skin Tone Evenness, Radiance/Brightness and Overall Healthy Appearance of Skin/Overall Skin Quality by using the Modified Griffith's Scale and its parameters of 0 = None (best possible outcome), 1-3 = Mild, 4-6 = Moderate, 7-9 = Severe (worst possible outcome). A decrease in scores indicates an improvement in study treatment efficacy. The null hypothesis is that the mean change from baseline is zero.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, MBA, Principal Investigator — Austin Institute for Clinical Research
Locations (1):
- Austin Institute for Clinical Research, Inc., Pflugerville, Texas, United States